CLINICAL TRIAL: NCT04275843
Title: The Effects of Western Diet Patterns on Plasma Inflammatory and Cardio Metabolic Health Signatures in Middle-aged Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: North Dakota Beef Commission (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: Pro00103827
Record Dates: First submitted 2020-02-07; First posted 2020-02-19 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-01

CONDITIONS: Healthy Diet

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: As this is feeding study with two very much different diets, participants and investigators were not blinded. The Core facilities that are analyzing de-identified coded samples and remain blinded to treatments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Diet (Active Comparator): Unprocessed/minimally processed whole foods.
  Interventions: Dietary Supplement: Traditional Diet
- Modern Diet (Active Comparator): Multi-ingredient, ultra-processed formulations of the traditional diet.
  Interventions: Dietary Supplement: Modern Diet

INTERVENTIONS:
Dietary Supplement: Traditional Diet — Consuming an traditional whole foods based diet for 4 weeks.
  Arms: Traditional Diet
Dietary Supplement: Modern Diet — Consuming an processed formulation of the traditional diet for 4 weeks.
  Arms: Modern Diet

SUMMARY:
The Western diet pattern or standard American diet is a modern dietary pattern that is characterized by high intakes of meat, pre-packaged foods, fried foods, high-fat dairy products, eggs, refined grains etc. When considering the role of saturated fat, it may be prudent to advise limiting all foods that contain saturated fats, including unprocessed/minimally processed meat, eggs, whole dairy in addition to processed, pre-packaged foods; however, this reductionist approach fails to take into account the food matrix and overall diet in which these nutrients are consumed.

Epidemiological evidence suggests that increased modern, pre-packaged food consumption is a major risk factor for metabolic disease by promoting inflammation. Based on these data, the investigators hypothesize that the pro-atherogenic effect of the Western diet is caused by the pro-inflammatory effects of consuming large amounts of modern ultra-processed foods, and that consumption of a similar amount of fat from minimally processed beef, poultry, dairy, eggs, as part of an unprocessed diet will positively impact inflammatory markers and lipoprotein profiles of study participants when compared to a diet rich in modern ultra-processed foods.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥35 and ≤60 years;
* BMI ≥25 and ≤35 kg/m2;
* Weight stable in last 3 months (Loss or gain <4%);
* Consistent physical activity levels;
* Hemoglobin A1C (HbA1C) ≤6.4%;
* Fasting insulin; <15 µU/mL;
* Fasting plasma glucose concentration <126 mg/dl;
* Willingness to eat the food provided in this study;
* Subjects must be able to speak and understand English to participate in this study
* Own a smartphone or other mobile device capable of downloading the Garmin Connect app.

Exclusion Criteria:

* Diagnoses of active malignancy, congestive heart failure, diabetes mellitus, chronic obstructive pulmonary disease, thyroid disease or other metabolic disorders that influence metabolism;
* Evidence of impaired kidney function (Estimated glomerular filtration rate [eGFR] <44 mL/min;
* Regular use of medication that interferes with the measurement of study outcomes as determined by the study team (e.g., NSAIDs, corticosteroids);
* Consuming >14 drinks per week of >4 drinks per night twice/week for male; >7 drinks per week or >3 drinks per night twice/week for female;
* Use of cigarettes (or other tobacco products) or use of any other (recreational) drug in last 3 months;
* Engaged in high-level competitive exercise (e.g., marathons, triathlons, cycling, weight-lifting competitions etc.)
* Self-reported sleep duration <5 hours per night;
* Any inflammatory diseases (e.g. asthma, autoimmune diseases, coeliac disease, glomerulonephritis, hepatitis, inflammatory bowel disease, arthritis);
* Use of antibiotics in last 30 days;
* Pregnant or lactating women;
* Eating disorders (e.g., anorexia nervosa, bulimia nervosa, binge eating disorders etc.)
* Psychological disorders (e.g., clinical depression, bipolar disorders etc.);
* Strict dietary patterns (e.g., vegan, carnivore, kosher, low-carb etc.);
* History of stomach or bowel resection (other than appendectomy), gastric bypass or other bariatric weight loss procedure effecting absorption;
* Persons who are not able to grant voluntary informed consent;
* Persons who are unable or unwilling to follow the study protocol or who, for any reason, the research team considers not an appropriate candidate for this study, including non-compliance with screening appointments or study visits.

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-12-21 (Actual); Study Completion 2021-12-21 (Actual)

PRIMARY OUTCOMES:
Change in plasma interleukin-6 levels | Baseline, up to 4 weeks.
  Plasma interleukin-6 levels will be measured before and after each diet
Change in plasma c-reactive protein levels | Baseline, up to 4 weeks.
  Plasma c-reactive protein levels levels will be measured before and after each diet
Change in plasma acylcarnitine profiles | Baseline, up to 4 weeks.
  Plasma acylcarnitines profiles levels will be measured before and after each diet

SECONDARY OUTCOMES:
Change in gut microbiota communities | Baseline, up to 4 weeks.
  Bifidobacterium, Faecalibacterium prausnitzii, Anerostipes, Roseburia
Energy expenditure | up to 4 weeks.
  Measured by the doubly labeled water method during the last week of each diet
Change in Neuroinflammation | Baseline, up to 4 weeks.
  Neurofilament light (NfL), glial fibrillary acidic protein (GFAP), Aß42 and p-tau will be measured before and after each diet

CONTACTS AND LOCATIONS:
Overall Officials: Stephan van Vliet, PhD, Study Director — Duke University; Kim Huffman, MD, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University School of Medicine, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No